CLINICAL TRIAL: NCT05171101
Title: The MAVEN Senior Scientist Initiative: A Trial of an Educational Training Program to Accelerate Diversity in Health & Science Leadership
Brief Title: The MAVEN Senior Scientist Initiative
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-0347
Record Dates: First submitted 2021-06-11; First posted 2021-12-28 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Lack of Diversity in Scientific Leadership
Keywords: Science; Scientists; Leadership; Women; Minority; Diversity; Virtual; Educational; Mentoring

STUDY DESIGN:
Intervention Model Description: Randomized Educational RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAVEN (Experimental)
  Interventions: Other: MAVEN
- Control (No Intervention): Participants enrolled in the control group will receive no mentoring activities but will complete all study measures and assessments.

INTERVENTIONS:
Other: MAVEN — The MAVEN education training program will be comprised of a 7-day virtual summer institute and a 7-day second virtual summer institute focused on respect-based leadership, senior scientist career planning, evidence-based mentoring, organizational culture problem solving, interdisciplinary team collaboration and inclusivity, effective science thought leadership, and public engagement. These summer institutes will be comprised of didactics, discussions, and interactive individual and team-based activities. Between the institutes there will be 10 months of mentorship, networking, and conduct of institutional change projects.
  Arms: MAVEN

SUMMARY:
MAVEN is an education training program designed to expand the national pool of qualified women and minority candidates for senior scientist positions across all NIGMS areas of science. Senior scientists (N=160, N=40 per cohort) belonging to an ethnicity, race or gender under-represented at the senior levels of faculty will be enrolled in a randomized 2-arm trial to determine the effects of the MAVEN intervention (comprised of virtual educational sessions and ongoing mentorship) on the following outcomes: 1) increased career satisfaction (primary outcome); 2) peak academic productivity; 3) expanded scientific networks; and 4) leadership ascension.

DETAILED DESCRIPTION:
The long-term objective of the MAVEN education training program is to expand the national pool of qualified women and minority candidates for senior scientist positions across all National Institute of General Medical Sciences (NIGMS) areas of science. The investigators intend to create a self-sustaining community committed to inclusive excellence in science. The investigators will do so by adapting best education practices from other industries in executive leadership, strategic career planning, and institution culture change, to create a sustainable, but intensive program with objective evaluation metrics. Using a randomized, 2-arm trial design, the investigators will enroll 40 senior scientists per year in 4 cohorts into the MAVEN study (160 participants total). Participants will be randomized to the MAVEN intervention group or the control group. Participants in the MAVEN group will receive two 7-day virtual institutes focused on senior scientist career planning, respect-based leadership, evidence-based mentoring, organizational culture problem solving, transparency and Open Science, interdisciplinary team collaboration and inclusivity, and effective science thought leadership. These summer institutes will be comprised of didactics, discussions, and interactive individual and team-based activities. Between the institutes there will be 10 months of mentorship, networking, and conduct of institutional change projects. Participants randomized to the control arm will complete all study measures but will not receive access to any of the virtual sessions or mentorship. Target program participants are scientists 10-15 years from their terminal degree , who identify as women, particularly as belonging to an ethnicity or race under-represented at the senior levels of faculty, and who currently hold one or more R01 or equivalent grants. To achieve the MAVEN long-term objective, scientists enrolled in the MAVEN intervention arm will be provided the skills to attain: 1) increased career satisfaction (primary outcome); 2) peak academic productivity; 3) expanded scientific networks; and 4) leadership ascension. Program success will be evaluated primarily by comparison of the control group to MAVEN scientists for change in career satisfaction scores, and also by a blended Major Educational Score Index comprised of h-index, relative citation ratio, number of publications in journals with an impact factor > 5, and annual federal grant dollar amounts. The investigators will also explore changes to professional scientific network size and the leadership ascension between the two groups, tested quantitatively. Primary, secondary, and exploratory outcomes will be evaluated at baseline for each cohort and yearly for all cohorts until the cessation of the program. If the scientific leaders and role models are diverse, the investigators of the current trial stand to benefit from enrichment of the pool of future investigators, the broader perspective in research agenda prioritization, the greater success in recruiting diverse research participants, and the enhanced ability to advance science to reduce health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Scientists 10 to 15 years from terminal degree in their field
* Identify as an ethnicity, race, or gender which is under-represented in senior levels of faculty.
* Have one or more funded R01 level grant (or equivalent level grant)

Exclusion Criteria:

* Scientists <10 or >15 years from terminal degree in their field
* Do not identify as an ethnicity, race, or gender which is under-represented in senior levels of faculty.
* Do not have one or more funded R01 level grant (or equivalent level grant)

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators will enroll participants who identify as women.
Enrollment: 160 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Career Satisfaction | Assessed at baseline and yearly afterwards until study completion 5 years following enrollment of the first cohort..
  Measured using the C-Change faculty satisfaction survey, a 74-item questionnaire assessing 12 areas including vitality, self-efficacy in career advancement, institutional support, relationships/inclusion/trust, values alignment, ethical/moral distress, respect, mentoring, leadership aspirations, work-life integration, gender equity, and equity for members of groups under-represented in medicine. Differences between the MAVEN and control groups will be assessed using a linear mixed model that includes an effect for treatment group, a fixed time effect, and group-time interaction, while accounting for within-subject correlation with a participant random effect. The investigators will use all observed data in an intent-to-treat manner. Investigators will also conduct GEE as a sensitivity analysis and each of the questions used in the survey will be summarized using proportions, and compared using Mann Whitney tests.

SECONDARY OUTCOMES:
Academic Productivity | Assessed at baseline and yearly afterwards until study completion 5 years following enrollment of the first cohort.
  Measured using the blended Major Educational Score Index (MESI). MESI will be a composite of four variables. First, the investigators will calculate the h-index from the Science Citation Index based on the number of peer-reviewed publications >h. Second, the investigators will compute the annual relative citation ratio, a quantitative assessment of scientific productivity, designed to assess the influence of a research article by considering its co-citation network and by field-normalizing that estimate. Third, the investigators will obtain the annual number of publications in journals with an impact factor 5 or above, and fourth, annual federal grant dollar amounts. MESI scores at program-end will be captured from various sources, standardized, and analyzed using linear mixed models, comparing the two groups with covariate adjustment. Detecting a significant difference between the MAVEN group and the control group at program-end would indicate success at attaining this objective.

OTHER OUTCOMES:
Professional Network Size | Assessed at baseline and yearly afterwards until study completion 5 years following enrollment of the first cohort.
  This will be assessed by co-authorship network analysis and content changes of the networks will be assessed by using natural language processing. Co-authorship network analysis measures trends in collaboration between scientists and identifies leaders in scientific fields. This is done by identifying manuscripts published by a participant, identifying the names and affiliations of all co-authors on those manuscripts, and using this information to construct an academic network around a particular participant. Change and expansion of the participant's network will be examined over time. The study team will calculate network measures and compare the structures between the MAVEN scholars and their control group over time. The investigators hypothesize a 5% greater expansion of scientific network size in the MAVEN group, relative to the comparison group at program-end.
Scientific Leadership Ascension | Assessed at baseline and yearly afterwards until study completion 5 years following enrollment of the first cohort.
  This will be assessed with an exploratory faculty title ascension analysis. Participant job titles will be obtained annually and will be classified by level of seniority with the input of the Advisory Committee. The study investigators will then code these titles, quantifying level of leadership ascension. The investigators will then conduct exploratory statistical analyses of the between-group differences in change in leadership across time.

CONTACTS AND LOCATIONS:
Overall Officials: Karina Davidson, PhD, MASc, Principal Investigator — Northwell Health
Locations (1):
- Institute of Health System Science, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be distributed. For program material deposit, the investigators will make all materials available from the MAVEN institute via the appropriate web internet repositories such as ABT, BEN Portal, MedEdPORTAL, NRMN, CTSA WIKI, NIH Distinguished Scholars Program, https://diversity.nih.gov/programs-partnerships/dsp, and other such entities. The trial pre-registration materials will be disseminated at Open Science and at clinicaltrials.gov. As stated in the Outcomes Data Collection and Storage Plan, all code, and data dictionaries and publications will be available in an Open Science framework. The investigators look forward to sharing curricula, group exercises, created case studies, other pedagogical materials, and evaluation plans and resulting data and findings with other diversity programs and with other training programs throughout the nation.